CLINICAL TRIAL: NCT04039893
Title: Prospective Trial to Evaluate MUltimodal Targeted Axillary Surgery (MUTAS) Approaches in Breast Cancer Patients With Positive Lymph Nodes.
Brief Title: MUltimodal Targeted Axillary Surgery
Acronym: MUTAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Collaborators: GEICAM (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/8361/I
Record Dates: First submitted 2019-06-19; First posted 2019-07-31 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Node-positive Breast Cancer
Keywords: axillary node clearance; axillary ultrasound imaging; sentinel node; tumor load
MeSH Terms: interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Node-positive breast cancer patients (Other): All patients with positive lymph nodes for who an axillary node clearance is proposed as part of the surgical treatment
  Interventions: Diagnostic Test: Systematic axillary ultrasound imaging; Diagnostic Test: Sentinel node; Procedure: Excision of suspicious lymph nodes; Procedure: Two steps axillary node clearance

INTERVENTIONS:
Diagnostic Test: Systematic axillary ultrasound imaging — Before surgery, all patients will be explored with a pre-defined systematic and reproducible axillary ultrasound imaging workflow intending to establish the number of neoplastic lymph nodes.
Diagnostic Test: Sentinel node — Sentinel nodes will be identified with a radioisotope tracer and blue dye or fluorescein.
Procedure: Excision of suspicious lymph nodes — Nodes suspected to be infiltrated both by physical exploration and/or ultrasound will be excised and evaluated separately.
Procedure: Two steps axillary node clearance — Axillary node clearance will be performed in two steps comprising inferior and superior clearance. The second intercostobrachial nerve will be considered the limit defining the border between superior and inferior axilla.

SUMMARY:
The present trial will prospectively evaluate the accuracy of both a systematic predefined axillary ultrasound imaging together with tumor load quantification of suspicious and sentinel axillary lymph nodes to predict overall tumor load in the axilla.

DETAILED DESCRIPTION:
Axillary node clearance (ANC) is a controversial intervention in the surgical treatment of breast cancer. Different studies have shown that in some patients with infiltrated axillary lymph nodes but low tumor burden, ANC can be safely omitted. However, indications for ANC persist in nowadays for patients with positive axillary lymph nodes and upfront surgery and patients with positive lymph nodes after neoadjuvant treatment. The present prospective study will evaluate the ability to establish an axillary tumor load with two steps. The first step will be a preoperative predefined systematic axillary ultrasound imaging workflow. The second step will be the tumor load evaluation of suspicious and sentinel axillary lymph nodes. We will also evaluate which patients have infiltrated nodes only beneath the second intercostobrachial nerve. The trial intends to identify patients for who a complete axillary node clearance could be spared.

ELIGIBILITY:
Inclusion Criteria:

* Node-positive breast cancer patients confirmed by biopsy or cytology
* Positivity confirmed before the surgical treatment

Exclusion Criteria:

* Inability to confirm positive lymph nodes by biopsy or cytology
* Inability to understand the protocol design
* Poor understanding of the Spanish language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2022-03-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients correctly identified as low axillary tumor load carriers by a pre-defined systematic axillary ultrasound imaging workflow | 24 months
  The accuracy (in terms of sensibility, specificity, positive predictive value and negative predictive value) of the pre-defined systematic ultrasound imaging workflow for identifying patients wih low axillary tumor load will be reported. Low axillary tumor load is defined as two or less infiltrated axillary lymph nodes.
Number of patients correctly identified as low axillary tumor load carriers by the information on tumor load of suspicious and sentinel axillary lymph nodes. | 24 months
  The accuracy (in terms of sensibility, specificity, positive predictive value and negative predictive value) of different tumor load cut-off points of the suspicious and sentinel axillary lymph nodes for identifying patients with low axillary tumor load will be reported.Low axillary tumor load is defined as two or less infiltrated axillary lymph nodes.
Number of patients correctly identified as low axillary tumor load carriers combining both the pre-defined axillary ultrasound imaging workflow with the information on tumor load of suspicious and sentinel axillary nodes | 24 months
  The accuracy (in terms of sensibility, specificity, positive predictive value and negative predictive value) of both the pre-defined systematic axillary ultrasound imaging workflow combined with tumor load information of suspicious and sentinel axillary lymph nodes for identifying patients with low axillary tumor load will be reported.Low axillary tumor load is defined as two or less infiltrated axillary lymph nodes.

SECONDARY OUTCOMES:
Number of infiltrated axillary lymph nodes detected by physical exploration | 24 months
  The difference between the number of positive lymph nodes identified in the final pathology exam and the nodes described as suspicious in physical exploration will be recorded to establish if physical exploration correctly estimates, underestimates or overestimates axillary tumour load.
Number of infiltrated lymph nodes detected by computed tomography | 24 months
  The difference between the number of positive lymph nodes identified in the final pathology exam and the nodes described as suspicious in computed tomography will be recorded to establish if physical exploration correctly estimates, underestimates or overestimates axillary tumour load.
Number of infiltrated lymph nodes detected by magnetic resonance | 24 months
  The difference between the number of positive lymph nodes identified in the final pathology exam and the nodes described as suspicious in magnetic resonance will be recorded to establish if magnetic resonance correctly estimates, underestimates or overestimates axillary tumour load.
Number of patients with low axillary tumor load among menopause status categories | 24 months
  The number of patients with low axillary tumor load in each menopause category will be reported. Patients will be categorized according to their menopausal status (pre-menopause and menopause).
Number of patients with low axillary tumor load among each breast cancer pathology subtype. | 24 months
  The number of patients with low axillary tumor load in each breast cancer pathology subtype (non-specified invasive carcinoma, lobular carcinoma and other carcinomas) will be reported
Number of patients with low axillary tumor load among each breast cancer immunophenotype. | 24 months
  The number of patients with low axillary tumor load in each breast cancer immunophenotypes (luminal , Her2 positive and triple negative carcinomas) will be reported
Number of patients with infiltrated nodes exclusively in the inferior axillary node clearance. | 24 months
  The number of patients with infiltrated nodes exclusively in the inferior axillary node clearance wil be reported. This information shall be obtained from the final pathology report.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vernet-Tomas, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernet-Tomas M, Banos N, Sabadell D, Corominas JM, Mestre-Fusco A, Suarez-Pinera M, Carreras R. p53 expression in breast cancer predicts tumors with low probability of non-sentinel nodes infiltration. J Obstet Gynaecol Res. 2015 Jul;41(7):1115-21. doi: 10.1111/jog.12670. Epub 2015 Feb 6. PMID 25657069
- [Background] Nicolau P, Gamero R, Rodriguez-Arana A, Plancarte F, Alcantara R, Carreras R, Sabadell D, Vernet-Tomas M. Imaging and pathology features to predict axillary tumor load in breast cancer. J Obstet Gynaecol Res. 2018 Feb;44(2):331-336. doi: 10.1111/jog.13490. Epub 2017 Oct 13. PMID 29027318